CLINICAL TRIAL: NCT01759446
Title: A Single-center, Randomized, Double-blind, Active- and Placebo Controlled, 5-way Crossover Study Assessing the Abuse Potential of Intranasally Administered VYCAVERT Tablets in Non-dependent Recreational Opioid Users.
Brief Title: Abuse Potential of Intranasal VYCAVERT Tablets (Hydrocodone Bitartrate/Acetaminophen) in Recreational Opioid Users
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acura Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AP-ADF-301
Record Dates: First submitted 2012-12-18; First posted 2013-01-03 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-08

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo taken first (Placebo Comparator): Placebo powder snorted with all other arms taken crossover therafter
  Interventions: Drug: Placebo taken first
- Generic H/A taken first (Active Comparator): Generic hydrocodone/APAP 10/325mg pulverized tablet snorted with all other arms taken crossover therafter
  Interventions: Drug: Generic H/A taken first
- Vycavert taken first (Active Comparator): Vycavert hydrocodone/APAP 10/325mg pulverized tablet snorted with all other arms taken crossover therafter
  Interventions: Drug: Vycavert taken first
- Generic H/A plus i taken first (Active Comparator): Generic hydrocodone/APAP 10/325mg plus additional inactive ingredients pulverized tablet snorted with all other arms taken crossover therafter
  Interventions: Drug: Generic H/A plus i taken first
- Generic H/A plus p taken first (Active Comparator): Generic hydrocodone/APAP 10/325mg plus one placebo pulverized tablet snorted with all other arms taken crossover therafter
  Interventions: Drug: Generic H/A plus p taken first

INTERVENTIONS:
Drug: Placebo taken first — Snorted in both nostrils within 5 minutes; 48 hours washout between doses
  Arms: Placebo taken first
Drug: Generic H/A taken first — Snorted in both nostrils within 5 minutes; 48 hours washout between doses
  Arms: Generic H/A taken first
Drug: Vycavert taken first — Snorted in both nostrils within 5 minutes; 48 hours washout between doses
  Arms: Vycavert taken first
Drug: Generic H/A plus i taken first — Snorted in both nostrils within 5 minutes; 48 hours washout between doses
  Arms: Generic H/A plus i taken first
Drug: Generic H/A plus p taken first — Snorted in both nostrils within 5 minutes; 48 hours washout between doses
  Arms: Generic H/A plus p taken first

SUMMARY:
To determine the relative abuse potential of VYCAVERT (hydrocodone bitartrate and acetaminophen) compared to GENERIC H/A (hydrocodone bitartrate and acetaminophen) when crushed and administered intranasally to non dependent, recreational opioid users.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests.
2. Subject is a recreational opioid user who is NOT dependent on opioids based on Diagnostic and Statistical Manual of Mental Disorders Fourth Edition Text Revision (DSM IV TR) criteria. A recreational opioid user is defined as a user of opioids for non medical purposes (i.e., for psychoactive effects) on at least 10 occasions within the last year and at least once in the 12 weeks before the Screening Visit (Visit 1).
3. Subjects must have experience with intranasal opioid administration, defined as intranasal use on at least 3 occasions within the last year before Screening.
4. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
5. Subject is able to speak, read, and understand English sufficiently to comprehend the nature of the study and to understand the informed consent form (ICF) and consent process.
6. An informed consent document signed and dated by the subject.
7. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

   -

Exclusion Criteria:

1. Diagnosis of substance and/or alcohol dependence (excluding caffeine and nicotine), as assessed by the Investigator using the DSM IV TR criteria.
2. Has participated in, is currently participating in, or is seeking treatment for substance and/or alcohol related disorders (excluding nicotine and caffeine).
3. Has a positive urine drug screen (UDS) including tetrahydrocannabinol (THC) at Screening (Visit 1). NOTE: Subjects with an opioid positive or THC-positive UDS at Visit 1 may be re tested once on or before Visit 2 (Day 0). If the UDS re test is negative, the subject can proceed to Visit 2. A positive UDS at Visit 2 will exclude the subject from further participation, unless the UDS is THC-positive in which the subject can continue in the study at the discretion of the Investigator.
4. Has a positive alcohol breath test at Screening. Positive results may be repeated and/or subjects re scheduled at the Investigator's discretion.
5. Has any condition in which an opioid is contraindicated (e.g., significant respiratory depression, acute or severe bronchial asthma or hypercarbia, suspected of having paralytic ileus).
6. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

   -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Webster, MD, Principal Investigator — Lifetree Clinical Research
Locations (1):
- Lifetree Clinical Research, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 44 recreational drug users with snorting experience were enrolled with 40 completing-Crossover designed
Pre-assignment Details: Each subject had to pass a blinded snorted drug discrimination phase to meet enrollment.
Groups:
- Placebo Taken First; Generic H/A Taken First; Vycavert Taken First; Generic H/A Plus i Taken First; Generic H/A Plus p Taken First: followed by all other drugs with 48 hours washout in between
Period: Overall Study
Arm/Group | Placebo Taken First | Generic H/A Taken First | Vycavert Taken First | Generic H/A Plus i Taken First | Generic H/A Plus p Taken First
Started | 9 | 9 | 9 | 9 | 8
Completed | 8 | 8 | 8 | 8 | 8
Not Completed | 1 | 1 | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Adult Recreational Snorting Drug Users who completed the study design per protocol
Groups:
- Placebo Taken First; Generic H/A Taken First; Vycavert Taken First; Generic H/A Plus i Taken First; Generic H/A Plus p Taken First: followed by all other doses crossover
- Total: Total of all reporting groups
Arm/Group | Placebo Taken First | Generic H/A Taken First | Vycavert Taken First | Generic H/A Plus i Taken First | Generic H/A Plus p Taken First | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 8 | 8 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.4 (3.99) | 24.4 (3.99) | 24.4 (3.99) | 24.4 (3.99) | 24.4 (3.99) | 24.4 (3.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 2 | 10
  Male | 6 | 6 | 6 | 6 | 6 | 30
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 8 | 40

OUTCOME MEASURES:

1. Primary Outcome: Emax - Maximum Drug Liking
Description: "Do you dislike or like the drug effect you are feeling now?" The question is scored using a 100-point bipolar visual analog scale (VAS) anchored in the center with "neither like nor dislike" (score of 50), on the left with "Strong Disliking" (score of 0) and on the right with "Strong Liking" (score of 100). Maximum Score. Assessment were made at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, and 8 hours post-dosing.
Time Frame: 8 hours
Population: Completers of all doses per protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Placebo
- Generic H/A; Vycavert: Hydrocodone and Acetaminophen
- Generic H/A Plus i: Hydrocodone/Acetaminophen with selected inactives
- Generic H/A Plus p: Hydrocodone/Acetaminophen plus placebo
Arm/Group | Placebo | Generic H/A | Vycavert | Generic H/A Plus i | Generic H/A Plus p
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40
score on a scale | 54.5 (8.52) | 75.0 (11.81) | 72.1 (12.98) | 75.6 (12.48) | 73.0 (13.13)

ADVERSE EVENTS:
Time Frame: AE's were collected as observed at systemically at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5 and 24 hours post-dose. AE's were observed and reported from first dose through the end of study (11 days).
Arm/Group | Placebo | Generic H/A | Vycavert | Generic H/A Plus i | Generic H/A Plus p
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44 | 0/44 | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44 | 0/44 | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 4/44 | 5/44 | 13/44 | 18/44 | 5/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | Generic H/A (N=44) | Vycavert (N=44) | Generic H/A Plus i (N=44) | Generic H/A Plus p (N=44)
Burning in throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (6) | 10 (10) | 3 (3) — Burning in nasal & throat
Nasal Burning (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 13 (13) | 18 (18) | 4 (4)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 5 (5) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No